CLINICAL TRIAL: NCT00005688
Title: Cardiac Arrhythmias and the Perception of Symptoms
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4184; R01HL043216 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac

SUMMARY:
To investigate the differential diagnosis and longitudinal course of medical outpatients complaining of palpitations. Also, to further examine the process of cardiac perception, the psychological factors which influence it, and the accurate awareness of cardiac arrhythmias.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

One hundred seventy-five consecutive patients referred for continuous ambulatory electrocardiographic (Holter) monitoring because of palpitations were studied. The investigators assessed cardiac symptoms, psychiatric diagnosis, life stress, beliefs about heart disease, somatization, and bodily absorption and amplification. Cardiac awareness, cardiac symptoms and cardiac activity were assessed during Holter monitoring and exercise tolerance testing (ETT). The referring physicians completed instruments rating their diagnostic impressions and clinical interventions. The patients' clinical course was then followed over the ensuing 12 months with telephone interviews and in-person assessments. These data permitted description and distinguished three subgroups of palpitation patients: those with panic disorder, in whom the symptom resulted from sympathetic nervous system arousal; those who were somatizing after a life event caused them to suspect that they had heart disease, in whom the palpitation resulted from a cognitive misattribution of benign bodily sensation; and those with clinically significant arrhythmias, whose symptoms resulted from a major cardiac irregularity. These findings were used to develop a clinical algorithm to aid in the differential diagnosis of palpitations and in identifying the patients most appropriate for Holter monitoring.

The patients' longitudinal course was followed to determine the predictors of continued somatization and chronicity, and to study their medical care by examining the referring physicians' diagnostic impressions and interventions. By comparing cardiac symptoms with concurrent cardiac activity during Holter monitoring and ETT, the investigators hoped to develop measures of cardiac awareness. They would then be able to describe inter-individual differences in cardiac awareness, examine several psychological factors which amplify or modulate awareness, and investigate the relationship between somatization and accuracy of symptom reporting. It was hoped that the findings would ultimately lead to improved cognitive and educational techniques to reassure and palliate palpitation patients, and to the early identification of patients who were unlikely to obtain symptomatic relief from antiarrhythmic therapy.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-07; Study Completion 1997-02 (Actual)

REFERENCES:
- [Background] Barsky AJ. A research agenda for outpatient consultation-liaison psychiatry. Gen Hosp Psychiatry. 1993 Nov;15(6):381-5. doi: 10.1016/0163-8343(93)90006-a. PMID 8112561
- [Background] Barsky AJ, Cleary PD, Brener J, Ruskin JN. The perception of cardiac activity in medical outpatients. Cardiology. 1993;83(5-6):304-15. doi: 10.1159/000175986. PMID 8111763
- [Background] Barsky AJ, Cleary PD, Coeytaux RR, Ruskin JN. The clinical course of palpitations in medical outpatients. Arch Intern Med. 1995 Sep 11;155(16):1782-8. PMID 7654112
- [Background] Barsky AJ, Ahern DK, Delamater BA, Clancy SA, Bailey ED. Differential diagnosis of palpitations. Preliminary development of a screening instrument. Arch Fam Med. 1997 May-Jun;6(3):241-5. doi: 10.1001/archfami.6.3.241. PMID 9161349
- [Background] Barsky AJ, Ahern DK, Bailey ED, Delamater BA. Predictors of persistent palpitations and continued medical utilization. J Fam Pract. 1996 May;42(5):465-72. PMID 8642363
- [Background] Barsky AJ, Delamater BA, Clancy SA, Antman EM, Ahern DK. Somatized psychiatric disorder presenting as palpitations. Arch Intern Med. 1996 May 27;156(10):1102-8. PMID 8638998
- [Background] Barsky AJ. Palpitations, cardiac awareness, and panic disorder. Am J Med. 1992 Jan 24;92(1A):31S-34S. doi: 10.1016/0002-9343(92)90134-w. PMID 1734732
- [Background] Barsky AJ, Cleary PD, Barnett MC, Christiansen CL, Ruskin JN. The accuracy of symptom reporting by patients complaining of palpitations. Am J Med. 1994 Sep;97(3):214-21. doi: 10.1016/0002-9343(94)90003-5. PMID 8092169
- [Background] Barsky AJ, Cleary PD, Coeytaux RR, Ruskin JN. Psychiatric disorders in medical outpatients complaining of palpitations. J Gen Intern Med. 1994 Jun;9(6):306-13. doi: 10.1007/BF02599176. PMID 8077994
- [Background] Barsky AJ, Cleary PD, Sarnie MK, Ruskin JN. Panic disorder, palpitations, and the awareness of cardiac activity. J Nerv Ment Dis. 1994 Feb;182(2):63-71. doi: 10.1097/00005053-199402000-00001. PMID 8308534
- [Background] Brown HD, Kosslyn SM, Delamater B, Fama J, Barsky AJ. Perceptual and memory biases for health-related information in hypochondriacal individuals. J Psychosom Res. 1999 Jul;47(1):67-78. doi: 10.1016/s0022-3999(99)00011-2. PMID 10511422
- [Background] Barsky AJ, Orav JE, Delamater BA, Clancy SA, Hartley LH. Cardiorespiratory symptoms in response to physiological arousal. Psychosom Med. 1998 Sep-Oct;60(5):604-9. doi: 10.1097/00006842-199809000-00016. PMID 9773765
- [Background] Barsky AJ, Ahern DK, Brener J, Surman OS, Ring C, Dec GW. Palpitations and cardiac awareness after heart transplantation. Psychosom Med. 1998 Sep-Oct;60(5):557-62. doi: 10.1097/00006842-199809000-00007. PMID 9773758
- [Background] Barsky AJ, Borus JF. Somatization and medicalization in the era of managed care. JAMA. 1995 Dec 27;274(24):1931-4. PMID 8568987